CLINICAL TRIAL: NCT03516682
Title: The REDIVAC Study-Reducing Delay in Vaccination of Children Study
Brief Title: Reducing Delay in Vaccination of Children: Logistic Barriers
Acronym: REDIVAC-LB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1R01HD079457 (NIH)
Record Dates: First submitted 2018-03-26; First posted 2018-05-04 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2018-08

CONDITIONS: Communicable Disease
Keywords: Logistic Barriers to Vaccination
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The Investigator and Analyst will stay blinded to the randomization arm throughout the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Parents will receive usual care for their child at Kaiser Permanente Colorado. This includes recommendations for well child visits at 2, 4, 6 and 12 months of age as well as automated reminders for age eligible children to receive the flu shot during flu season.
- Reminders (Experimental): Parents randomized to the reminder arm will receive automated reminders to complete a 6 month and 12 month vaccine visit for their child. They will receive 2 reminders before the child is 6 and 12 months of age and 2 reminders after their child is 6 and 12 months of age. Reminders will not occur if they have received vaccines within the eligible time frame to receive a vaccine or have a visit scheduled. After randomization, participants in the intervention arm will have an opportunity to provide their preference on how they receive reminders (text, phone and/or email). Participants not providing a preference will receive text reminders. If a child is randomized into the study after the child is 7 months of age, the parent will only be eligible for reminders for the 12 month vaccine visit.
  Interventions: Behavioral: Reminders

INTERVENTIONS:
Behavioral: Reminders — Automated reminders for the 6 month and 12 month vaccine visits for parents experiencing logistic barriers to vaccination.
  Other Names: REDIVAC-Logistic Barriers
  Arms: Reminders

SUMMARY:
This study will assess the impact of automated reminders for the 6 month and 12 month vaccine visits to increase vaccination in parents experiencing logistic barriers to vaccination.

DETAILED DESCRIPTION:
Parents of children less than 11 months of age will be identified as delayed or missing vaccinations due to logistic barriers in the Kaiser Permanente Colorado population. Parents identified will be randomized to the intervention arm or the usual care arm. Those in the intervention arm will receive automated reminders for the 6 month and 12 month vaccine visits. Reminders will include scheduling information as well as access to a website with vaccine and scheduling information. They will also have an opportunity to provide preferences in how they receive the automated reminders (text, phone or email). There will be 2 reminders before the 6 and 12 month visits and 2 after the 6 and 12 month visits. Parents will be excluded from receiving reminders if they have received vaccines within the time frame when they are eligible to receive another vaccine or have a well child visit scheduled.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children less than 11 months of age
* Currently enrolled at Kaiser Permanente Colorado at the time of identification
* The child is missing recommended vaccinations

Exclusion Criteria:

* Non-english speaking
* diagnosis code indicating parent vaccine refusal

Ages: 1 Month to 11 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Vaccines received (Electronic Health Record) | up to a year of follow up
  Vaccination records from the participants electronic health record will be used to measure vaccines received. Vaccines received is a dichotomous variable indicating if any vaccines were received while enrolled in the study

SECONDARY OUTCOMES:
Vaccine dose (Electronic Health Record) | up to a year of follow up
  Vaccination records from the participants electronic health record will be used to measure vaccine dose. Vaccine dose is a measure of the vaccine doses that the child could have received while enrolled in the study, the number of vaccine doses received

CONTACTS AND LOCATIONS:
Overall Officials: Jason Glanz, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Colorado Institute for Health Research, Denver, Colorado, United States

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276